CLINICAL TRIAL: NCT03412370
Title: Symptom Tracking in Women Following Mammography
Brief Title: Questionnaires and Cognitive Assessments Following Mammography
Status: Terminated | Type: Observational
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-17-2; NCI-2017-02234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-17-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Health Status Unknown
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires, cognitive assessment): Patients complete questionnaires and cognitive assessments over 45-60 minutes within 3 weeks following mammography and at about 3 months in patients for whom biopsy is not required, before biopsy and at about 3 months in patients for whom biopsy is required, and at 4-6 weeks after first chemotherapy infusion in patients receiving chemotherapy.
  Interventions: Other: Cognitive Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cognitive Assessment — Complete cognitive assessments
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This pilot research trial studies how well questionnaires and cognitive assessments work in tracking patient symptoms following mammography. Gathering information over time through questionnaires and cognitive tests about symptoms patients may experience after a mammogram may help doctors understand the cause of these symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of Internet-based cognitive assessments as preliminary data prior to larger clinical trial.

OUTLINE:

Patients complete questionnaires and cognitive assessments over 45-60 minutes within 3 weeks following mammography and at about 3 months in patients for whom biopsy is not required, before biopsy and at about 3 months in patients for whom biopsy is required, and at 4-6 weeks after first chemotherapy infusion in patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Mammography Breast Imaging Reporting and Data System (BI-RAD) 4-5; or BI-RAD 1-2
* Fluent in English
* Access to Internet
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Prior abnormal mammography
* Prior cancer diagnosis
* Prior treatment with chemotherapy

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who have just completed a mammography
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Number of patients invited who agree to participate | Up to 2 years
  Number of patients invited will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Broderick, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States